CLINICAL TRIAL: NCT05635526
Title: Assessment of Corneal Biomechanics With the Corvis ST in Different Age of Myopia With Orthokeratology
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022049
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-10

CONDITIONS: Myopia; Orthokeratology
Keywords: Myopia prevention and control; Orthokeratology; Dynamic corneal response
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: 8-12 years old
- 2: 13-16 years old
- 3: over 16 years old

SUMMARY:
The present research focused on the effect of the age for the corneal biomechanics of low and moderate myopia patients after wearing orthokeratology (OK lens). According to age, the included cases were divided into 3 groups. Through the analysis of corneal biomechanical parameters, further learn the influence of OK lens on the patient cornea. It would help ophthalmologist and optometrist find out the potential issue and reach a better control result.

DETAILED DESCRIPTION:
The present research focused on the effect of the age for the corneal biomechanics of low and moderate myopia patients after wearing orthokeratology (OK lens). According to age, the included cases were divided into 3 groups: Ⅰ (8-12 years old), Ⅱ (13-16 years old), Ⅲ (over 16 years old). The OK lenses used in the present study are of the same design (Euclid Systems Orthokeratology; Euclid System, Herndon, VA, USA). The base line (Day 0) and different follow-up time point (Day 1, Week 1, Week 2, Month 1, Month 3, and Month 6) of dynamic corneal response (DCR) (including 19 items) of the patients derived by Corvis ST were collected. The difference between before and after wearing OK Lens and the changes of parameters among the three groups were both analyzed. And the correlation between axis length (AL) and the 19 parameters also was analyzed. Through the analysis of corneal biomechanical parameters, further learn the influence of OK lens on the patient cornea. It would help ophthalmologist and optometrist find out the potential issue and reach a better control result.

ELIGIBILITY:
Inclusion Criteria:

* age from 8 to 40 years old
* spherical equivalent(SE) was range from -1.00D to -5.00D
* conform to the standard of wearing orthokeratology lens

Exclusion Criteria:

* ocular diseases and systemic diseases
* visual acuity was less than 20/20
* unable to follow visitors on time

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Myopia with orthokeratology lens and complete follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
The change of dynamic corneal response (DCR) | The change of baseline and 1 day, 1 week, 2 weeks, 1 month, 3 months, and 6 months
  The axial length was measured by Corvis ST

SECONDARY OUTCOMES:
The change of axial length | The change of baseline and 6 months
  The axial length was measured by AL-scan

CONTACTS AND LOCATIONS:
Locations (1):
- Tiajin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No